CLINICAL TRIAL: NCT00984334
Title: A Multicentre, Randomised, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study Evaluating the Safety, Tolerability and Efficacy of Naloxone SR Capsules in Subjects With Constipation Due to Opioids, Taken for Persistent Non-Cancer Pain
Brief Title: Naloxone SR Capsules in Patients With Opioid Induced Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAL-OIC-01; 2009-009377-10 (EudraCT Number)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Pain; Opioid Induced Constipation
Keywords: pain; opioid; constipation; Subjects taking opioids for chronic non-cancer pain, who; experience symptoms of opioid induced constipation
MeSH Terms: conditions — Chronic Pain; Opioid-Induced Constipation; Pain; Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Capsules with no active drug (Placebo Comparator): Placebo capsules once daily for three weeks then twice daily for three weeks.
  Interventions: Drug: Placebo
- Naloxone SR 2.5 mg capsules (Active Comparator): Naloxone SR 2.5 mg capsules once daily for three weeks then twice daily for three weeks.
  Interventions: Drug: Naloxone SR 2.5 mg capsules
- Naloxone SR 10mg capsules (Experimental): Naloxone SR 10 mg capsules once daily for three weeks then twice daily for three weeks.
  Interventions: Drug: Naloxone SR 10 mg capsules
- Naloxone SR 20 mg capsules (Experimental): Two Naloxone SR 10 mg capsules once daily for three weeks then twice daily for three weeks.
  Interventions: Drug: Naloxone SR 20mg capsules
- Naloxone SR 5mg capsules (Experimental): Naloxone SR 5 mg capsules once daily for three weeks then twice daily for three weeks.
  Interventions: Drug: Naloxone SR 5 mg capsules

INTERVENTIONS:
Drug: Naloxone SR 5 mg capsules
  Arms: Naloxone SR 5mg capsules
Drug: Placebo
  Arms: Capsules with no active drug
Drug: Naloxone SR 10 mg capsules
  Arms: Naloxone SR 10mg capsules
Drug: Naloxone SR 20mg capsules
  Arms: Naloxone SR 20 mg capsules
Drug: Naloxone SR 2.5 mg capsules
  Arms: Naloxone SR 2.5 mg capsules

SUMMARY:
For many patients taking opioids for pain relief one of the most distressing side effects is constipation. Naloxone is effective in the reversal of the effects of opioids and is used following opioid overdose. If naloxone is given by mouth it would relieve the effects of constipation but as it goes into the blood stream very quickly, it would also reverse the effects of the opioid and therefore stop the pain relief. The aim of this study is to examine a slow release formulation of naloxone to see if is can reduce constipation without reducing the pain relieving effects of the opioid.

DETAILED DESCRIPTION:
Naloxone has been used for many years as an IV or IM injection for the reversal of opioid effects (following opioid overdose) and has been evaluated as an oral formulation to manage opioid-induced constipation. Immediate release oral naloxone preparations have however led to reversal of opioid effects and withdrawal. This has initiated the development of prolonged (slow release) naloxone preparations which prevent the systemic levels of naloxone reaching levels where the central opioid effects may be reversed. Naloxone has a high first pass metabolism (98%) and short half life (~1hr).

The objectives of this trial are to identify the optimum dosage regime of Naloxone SR capsules based on tolerability level, to improve spontaneous bowel movement frequency, and relieve GI symptoms, in patients suffering with opioid induced constipation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must give written informed consent
* Male or female subjects greater than 18 years of age
* Taking opioid full agonist therapy(oral or transdermal) for persistent non-cancer pain, for at least 4 weeks prior to baseline visit
* Subjects with at least a 3 week history of OIC prior to baseline; where bowel dysfunction is predominantly due to opioids and started following commencement of opioid therapy
* Subjects with <3 SBMs a week and experiencing one or more bowel symptoms (incomplete evacuation, straining, hard/small pellets) for 25% or more of bowel movements during the screening period
* Subjects must be willing to discontinue all current laxative (constipation) therapy. Bisacodyl will be provided and taken as required

Exclusion Criteria:

* Women of childbearing potential, unless surgically sterile or using adequate contraception (either IUD, oral or depot contraceptive, or barrier plus spermicide). Women using oral contraception must have started using it at least 2 months prior to enrolment
* Women who are pregnant or breastfeeding
* Symptoms suggestive of non-opioid related bowel dysfunction (e.g. IBS - intermittent constipation or diarrhoea) or have diarrhoea or loose stools in the 4 weeks prior to baseline
* History of chronic constipation prior to commencing opioid therapy
* Gastrointestinal disorders known to affect bowel transit, or contribute to bowel dysfunction (other than OIC)
* Chronic faecal incontinence
* Subjects who have a colostomy, ileostomy, or colectomy with ileorectal anastomosis
* Subjects with a history of neoplastic disease within 5 years (except for basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin)
* Subjects taking opioids for the management of drug addiction Subjects who do not meet any of the following criteria regarding baseline medications. Analgesia (including opioids and NSAIDs) should be stable throughout the trial.

  * Any baseline analgesia must have been administered at a stable dose for a minimum of 4 weeks. If non-opioid analgesia recently discontinued, must have stopped at least 4 weeks prior to baseline
  * Laxatives (outside that allowed by the protocol) are not permitted; these agents must have been discontinued at the screening visit.
  * Use of drugs known to affect gut transit time (other than opioids) are not permitted (see Section 6.9 for exceptions)
  * Use of mixed agonist/antagonist, or partial agonist opioids are not permitted (e.g. buprenorphine, pentazocine, cyclazocine, nalbuphine, nalorphine)
  * Experimental agents must have been discontinued at least 8 weeks prior to screening, or for a period equivalent to 5 half-lives (t½) of the agent (whichever is longer)
  * Subjects with a history of clinically significant and/or persistent disorder that, in the investigators opinion, may affect the clinical trial assessments
  * Subjects with any laboratory tests considered clinically significant at screening.
  * Subjects not ambulatory i.e. bedridden or require use of a commode
  * Subjects who will be unavailable for the duration of the trial, likely to be non-compliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Simpson, MD, Principal Investigator — St James University Hospital, Leeds, UK
Locations (8):
- Germany (5):
  - Schmerzzentrum Berlin, Berlin
  - Schmerzzentrum Frankfurt, Frankfurt
  - Gemeinschaftspraxis Tamm-Albert-Schroter-Uhmann, Hanover
  - Gemeinschaftspraxis Loewenstein-Hesselbarth, Mainz
  - Regionales Schmerzzentrum Wuppertal, Wuppertal
- United Kingdom (3):
  - St Jame's Hospital Leeds, Leeds
  - Norfolk & Norwich Hospital, Norwich
  - Department of Pain Management, York Hospital, York

RESULTS

PARTICIPANT FLOW:
Groups:
- Capsules With no Active Drug: Placebo capsules once daily for three weeks then twice daily for three weeks.
  Placebo :
- Naloxone SR 10mg Capsules: Naloxone SR 10 mg capsules once daily for three weeks then twice daily for three weeks.
  Naloxone SR 10 mg capsules :
- Naloxone SR 2.5 mg Capsules: Naloxone SR 2.5 mg capsules once daily for three weeks then twice daily for three weeks.
  Naloxone SR 2.5 mg capsules :
- Naloxone SR 20 mg Capsules: Two Naloxone SR 10 mg capsules once daily for three weeks then twice daily for three weeks.
  Naloxone SR 20mg capsules :
- Naloxone SR 5mg Capsules: Naloxone SR 5 mg capsules once daily for three weeks then twice daily for three weeks.
  Naloxone SR 5 mg capsules :
Period: Overall Study
Arm/Group | Capsules With no Active Drug | Naloxone SR 10mg Capsules | Naloxone SR 2.5 mg Capsules | Naloxone SR 20 mg Capsules | Naloxone SR 5mg Capsules
Started | 8 | 8 | 8 | 8 | 8
Completed | 7 | 7 | 8 | 7 | 7
Not Completed | 1 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capsules With no Active Drug | Naloxone SR 10mg Capsules | Naloxone SR 2.5 mg Capsules | Naloxone SR 20 mg Capsules | Naloxone SR 5mg Capsules | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 7 | 8 | 7 | 35
  >=65 years | 1 | 2 | 1 | 0 | 1 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.2) | 53.4 (15.7) | 50.6 (12.7) | 48.6 (8.6) | 60.5 (8.8) | 53.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 1 | 5 | 21
  Male | 2 | 3 | 4 | 7 | 3 | 19
Region of Enrollment [Number; unit: participants]
  Germany | 5 | 6 | 2 | 5 | 8 | 26
  United Kingdom | 3 | 2 | 6 | 3 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment Emergent Adverse Events on Single Dosing.
Description: Incidence and severity of treatment emergent adverse events on single dosing.
Time Frame: 3 weeks
Population: Intent to treat.
Measure: Number; unit: participants
Arm/Group | Capsules With no Active Drug | Naloxone SR 10mg Capsules | Naloxone SR 2.5 mg Capsules | Naloxone SR 20 mg Capsules | Naloxone SR 5mg Capsules
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
participants | 8 | 5 | 4 | 6 | 6

ADVERSE EVENTS:
Arm/Group | Capsules With no Active Drug | Naloxone SR 10mg Capsules | Naloxone SR 2.5 mg Capsules | Naloxone SR 20 mg Capsules | Naloxone SR 5mg Capsules
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 5/8 | 5/8 | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsules With no Active Drug (N=8) | Naloxone SR 10mg Capsules (N=8) | Naloxone SR 2.5 mg Capsules (N=8) | Naloxone SR 20 mg Capsules (N=8) | Naloxone SR 5mg Capsules (N=8)
Panic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — panic attack during pre-treatment screening phase.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsules With no Active Drug (N=8) | Naloxone SR 10mg Capsules (N=8) | Naloxone SR 2.5 mg Capsules (N=8) | Naloxone SR 20 mg Capsules (N=8) | Naloxone SR 5mg Capsules (N=8)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (25) | 4 (14) | 2 (3) | 3 (10) | 3 (3)
General disorders and administration site conditions (General disorders) | 3 (3) | 2 (3) | 1 (1) | 2 (2) | 3 (4)
Nervous system disorders (Nervous system disorders) | 1 (1) | 2 (5) | 2 (2) | 4 (8) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects per group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less